CLINICAL TRIAL: NCT02859909
Title: An Open Label, Prospective, Randomized, Multicenter Study Investigating Clinical Efficacy and Safety of the Human Normal Immunoglobulin for Intravenous Administration BT595 in Patients With Chronic Primary Immune Thrombocytopenia (ITP)
Brief Title: This Clinical Study is to Test Efficacy and Safety of BT595 in Chronic Primary Immune Thrombocytopenia (ITP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotest (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 992
Record Dates: First submitted 2016-07-25; First posted 2016-08-09 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2018-04

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 day treatment schedule (Experimental): Patients will receive a dosage of 1 g/kg bw per day of BT595 for 2 consecutive days
  Interventions: Biological: BT595
- 5 day treatment schedule (Experimental): Patients will receive a dosage of 0.4 g/kg bw per day of BT595 for 5 consecutive days
  Interventions: Biological: BT595

INTERVENTIONS:
Biological: BT595
  Other Names: Human Immunoglobulin

SUMMARY:
The main purpose of this study is to assess the efficacy and safety of BT595 in adult subjects with chronic ITP. The primary objective of this study is to determine the rate of subjects with a response. A response is defined as a platelet count of ≥30×10^9/L and at least a 2 fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart, and the absence of bleeding. The secondary objectives of this study, in addition to further efficacy assessments, are to evaluate the safety of BT595.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of chronic ITP (>12 months' duration), including diagnosis of refractory ITP, and as defined by the International Working Group (Rodeghiero et al, 2009), where ITP is described as an autoimmune disorder characterized by isolated thrombocytopenia in the absence of other causes or disorders that may be associated with thrombocytopenia
* Treatment is indicated because of a high risk of bleeding or a need to raise the platelet count
* Mean screening platelet count of <30×10^9/L from 3 qualifying platelet counts performed within approximately 7 to 14 days before the start of treatment, with no individual platelet count above 35×10^9/L. The subject may be rescreened if the mean screening platelet count is ≥30×10^9/L. (Note: If a subject is rescreened, all screening laboratory tests must be repeated.)

Main Exclusion Criteria:

* Secondary thrombocytopenia or acquired medical conditions known to be associated with secondary thrombocytopenia, such as chronic lymphocytic leukemia; lymphoma; multiple myeloma; thyroid disease; or other forms of thrombocytopenia, such as drug induced thrombocytopenia; cirrhotic liver diseases; antiphospholipid syndrome; environmental thrombocytopenia; and bone marrow diseases
* Severe concomitant diseases that in the judgment of the investigator will interfere with the study, such as autoimmune hemolytic anemia, acute renal failure, and noncontrolled arterial hypertension
* Laboratory findings (e.g., abnormal laboratory values for hemoglobin, transaminase levels [alanine aminotransferase, aspartate aminotransferase], total bilirubin, creatinine, blood urea nitrogen, and immunoglobulins G, A, M) that preclude participation
* Positive Coombs test (direct and indirect)
* Planned invasive procedures during the time frame of the study
* Maintenance therapy with intravenous immunoglobulins (IVIgs) or infusion of IVIgs within 3 months before start of the study
* Unresponsive to previous IVIg treatment
* Additional therapy with high dose corticosteroids (equivalent to >30 mg prednisone/day), thrombopoietin receptor agonists, and/or immunosuppressives and/or other therapies (e.g., infusion of platelets) within 1 month before the start of the study (Note: Subjects on stable doses of ITP active treatment must not have modified the dose in the preceding 2 weeks and must maintain their prestudy dose during the study. Corticosteroids should not be given as a premedication. Rescue therapy with short courses [i.e., 1 to 4 days] of high dose steroids and IVIgs are allowed up to 2 weeks before study inclusion.)
* History of thrombotic events (including myocardial infarction, cerebral vascular accident [including stroke], pulmonary embolism, and deep vein thrombosis) 6 months before treatment start with BT595 or the presence of significant risk factors for thrombotic events
* Therapy with live attenuated virus vaccines 3 months before start of the study
* Selective, absolute immunoglobulin A (IgA) deficiency or known antibodies to IgA

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Rate of subjects with response (R) | 1 month
  The rate of subjects with response is defined as subjects with a platelet count of ≥30×10^9/L and at least a 2 fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart, and the absence of bleeding

SECONDARY OUTCOMES:
The number of subjects with complete response (CR) | 1 month
  The number of subjects with CR, which is defined as a platelet count ≥100×10^9/L, confirmed on at least 2 separate occasions at least 7 days apart, and the absence of bleeding
The percentage of subjects with complete response (CR) | 1 month
  The percentage of subjects with CR, which is defined as a platelet count ≥100×10^9/L, confirmed on at least 2 separate occasions at least 7 days apart, and the absence of bleeding
The number of subjects with no response (NR) | 1 month
  The number of subjects with NR, which is defined as subjects without R, i.e. a platelet count <30×10^9/L or less than a 2 fold increase of baseline platelet count, confirmed on at least 2 separate occasions, approximately 1 day apart, or bleeding
The percentage of subjects with no response (NR) | 1 month
  The percentage of subjects with NR, which is defined as subjects without R, i.e. a platelet count <30×10^9/L or less than a 2 fold increase of baseline platelet count, confirmed on at least 2 separate occasions, approximately 1 day apart, or bleeding
The number of subjects with a loss of response | 1 month
  The number of subjects with a loss of response (only in subjects who previously had CR or R), which is defined as a platelet count <100×10^9/L or bleeding (from CR) or platelet count <30×10^9/L or less than 2 fold increase of the baseline platelet count, or bleeding (from R). Platelet counts will be confirmed on at least 2 separate occasions approximately 1 day apart
The percentage of subjects with a loss of response | 1 month
  The percentage of subjects with a loss of response (only in subjects who previously had CR or R), which is defined as a platelet count <100×10^9/L or bleeding (from CR) or platelet count <30×10^9/L or less than 2 fold increase of the baseline platelet count, or bleeding (from R). Platelet counts will be confirmed on at least 2 separate occasions approximately 1 day apart
Time to Response (R) | 1 month
  Time to response (R), which is defined as the time from the start of treatment to the time of achievement of CR or R
Duration of response (R), | 1 month
  Duration of response (R), which is defined as the time from the achievement of CR or R to loss of CR or R
The number of subjects with response to ≥50×10^9/L | 1 month
  The number of subjects with response to ≥50×10^9/L, which is defined as a platelet count increase to at least ≥50×10^9/L within 7 days of the first BT595 infusion
The percentage of subjects with response to ≥50×10^9/L | 1 month
  The percentage of subjects with response to ≥50×10^9/L, which is defined as a platelet count increase to at least ≥50×10^9/L within 7 days of the first BT595 infusion
Subject's maximum platelet count achieved | 1 month
Time to subject's maximum platelet count | 1 month
Time course of platelet count | 1 month
Occurrence of bleeding symptoms | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Judit Demeter, MD, PhD, DSc, Principal Investigator — Semmelweis University Medical School, First Department of Medicine, Department of Hematology, 1083 Budapest, Korányi S. u. 2/a, Hungary
Locations (22):
- Bulgaria (5):
  - Investigational site # 3597, Pleven
  - Investigational site # 3593, Plovdiv
  - Investigational site # 3598, Sofia
  - Investigational site # 3591, Sofia
  - Investigational site # 3596, Varna
- Investigational site # 4202, Prague, Czechia
- Germany (2):
  - Investigational site # 4901, Berlin
  - Investigational Site #4902, München
- Hungary (6):
  - Investigational site # 3601, Budapest
  - Investigational site # 3604, Debrecen
  - Investigational site # 3607, Győr
  - Investigational site # 3602, Miskolc
  - Investigational site # 3603, Nyíregyháza
  - Investigational site # 3606, Pécs
- Serbia (4):
  - Investigational site # 3811, Belgrade
  - Investigational site # 3813, Belgrade
  - Investigational site #3814, Niš
  - Investigational site # 3812, Novi Sad
- Spain (4):
  - Investigational site # 3403, Madrid
  - Investigational site # 3404, Madrid
  - Investigational site #3401, Málaga
  - Investigational site # 3402, Palma de Mallorca

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demeter J, Hamed A, Laszlo S, Suvajdzic N, Aigner S, Borner B, Staiger C. Efficacy and safety of BT595 (10% human intravenous immunoglobulin) in adult patients with chronic immune thrombocytopenia. Transfus Med. 2023 Apr;33(2):165-173. doi: 10.1111/tme.12943. Epub 2022 Nov 30. PMID 36448274